CLINICAL TRIAL: NCT05687513
Title: Clinical Efficacy and Mechanism of Yisui Granule in Treatment of Low and Medium Risk Myelodysplastic Syndrome Through Demethylation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Wang Jing, associate professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-09-01
Record Dates: First submitted 2022-10-30; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: MDS

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental)
  Interventions: Drug: Yisui granule
- control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Yisui granule — Yisui granule
  Arms: treatment group
Drug: Placebo — placebo
  Arms: control group

SUMMARY:
The goal of this clinical trial is to explore the mechanism of Yisui Granule(YSG) in the treatment of myelodysplastic syndrome(MDS) through demethylation.

Under the same condition of basic western medicine treatment, the treatment group used the same traditional Chinese medicine decoction pieces as YSG, and the control group was given placebo. Through a randomized controlled clinical study, we focused on observing the effects of MDS patients on clinical symptoms (including single symptom), fatigue relief, quality of life, peripheral blood picture, blood transfusion interval and blood transfusion volume, and measured the expression of DNMTs, the expression and methylation level of Wnt3a、β-catenin、SFRP and other indicators, as well as cytokines, were used to explore the mechanism of YSG in the treatment of MDS through demethylation.

ELIGIBILITY:
A. Diagnosed as myelodysplastic syndrome, IPSS score 0-1; B. It meets the syndrome standard of "deficiency of both qi and yin, internal resistance of blood stasis"; C. Newly diagnosed cases or no application of other Chinese and western medicines or treatment schemes in the past month; D. Take the test voluntarily and sign the informed consent form.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Methylation index | 8 weeks

IPD SHARING:
Plan to Share IPD: No